CLINICAL TRIAL: NCT05019144
Title: A Novel Telemedicine Optimized Burn Intervention (TOBI) for Pediatric Burn-injured Patients and Their Caregivers
Brief Title: Telemedicine Optimized Burn Intervention
Acronym: TOBI
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Medical University of South Carolina (Other)
Collaborators: Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Diagnostic
Other Study IDs: Pro00109037; K23HD098328-01A1 (NIH)
Record Dates: First submitted 2021-08-18; First posted 2021-08-24 (Actual); Results first posted 2025-07-11 (Actual); Last update posted 2025-07-11 (Actual); Status verified 2025-06

CONDITIONS: Burns; Pediatric ALL
Keywords: Pediatrics; Telemedicine; Mobile health; Burns
MeSH Terms: conditions — Burns; Precursor Cell Lymphoblastic Leukemia-Lymphoma

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Face-to-face arm (Active Comparator): Standard face-to-face burn care.
  Interventions: Procedure: Face-to-face burn care
- TOBI arm (Experimental): A novel smartphone application for burn wound care, called the Telemedicine Optimized Burn Intervention (TOBI), was recently developed to enable burn experts to direct burn wound care while the patient and caregiver are home through text messaging and video-conferencing. The app was designed to bring expert wound care directly to the patient's home to address barriers to healthcare, including high cost burden and time commitment (e.g., geographic limitations, transportation to burn centers, parking, lodging, meals, time away from school and work), particularly for patients/families in rural and medically underserved communities. TOBI is synced with a portal used by providers, as an adjunct to standard therapy. This burn app provides education through frequently asked questions, instructional burn dressing change videos in addition to direct communication between patient and burn expert through store-and-forward pictures and videoconferencing.
  Interventions: Procedure: Telemedicine enhanced burn care

INTERVENTIONS:
Procedure: Face-to-face burn care — If the participants are assigned to FTF care, they will receive standard burn care including a return follow-up in the burn clinic on a routine basis as prescribed by the clinical burn team (at least once per week) until the burn has healed.
  Arms: Face-to-face arm
Procedure: Telemedicine enhanced burn care — Participants assigned to TOBI will be given instructions how to download and use TOBI on a smartphone, including how to interface with burn clinicians using text-messaging, videoconferencing, and sending photos of the child's burn(s). The participants will have scheduled video visits with the care provider at least weekly until the burn has healed. The participants will be able to use other features of the app, such as text-messaging and sending photos of the burn(s), as needed. The participants will be able to use standard FTF burn care as well. They will be given instructions how to contact the burn team through the hospital paging operator if TOBI is unavailable or there is an emergency.
  Arms: TOBI arm

SUMMARY:
Because burn patients and their caregivers often live long distances from regional burn centers, access to expert burn care is limited, resulting in a negative effect on adherence to treatment and a higher risk of wound complication. A novel smartphone application synchronized with a web portal for providers, called the Telemedicine Optimized Burn Intervention (TOBI), was recently developed to enable burn experts to direct burn wound care while the patient and caregiver are home through text messaging, image transfer, and video-conferencing. The goal of the present study is evaluate TOBI compared to face-to-face care as usual for pediatric patients/caregivers visiting a burn center. This study will also assess the feasibility of conducting a larger-scale clinical trial in several burn centers. The app will allow the physician and patient/caregivers to make instant decisions regarding treatment, allowing for "turn on a dime" treatment decisions, rather than having the patients and families wait for scheduled clinic appointments, often hours away from home. This "on demand" medical care takes an innovative approach to increasing access to burn experts through smartphone technology and addressing adherence to prescribed treatment by increasing communication between provider and patients.

ELIGIBILITY:
Inclusion criteria:

Caregiver parents and their children (patients) will be considered as participants and will be eligible for enrollment if:

1. the patient (child) is < 18 years of age; caregiver age >18 years of age
2. the patient is diagnosed with a partial thickness burn between <1% TBSA - 20% TBSA by a pediatric burn surgeon;
3. the patient's burn is being treated with advanced burn dressing therapy (e.g., Silvadene™, Polysporin™, Acticoat™, Mepilex™, or Mepitel™);
4. the patient's burn is evaluated by the MUSC burn team within 48 hours of injury;
5. the patient's caregiver (parent or legal guardian) is able to speak, hear, and understand English, as determined during study recruitment procedures;
6. the caregiver owns and is capable of using a smart device (an Android or iOS smartphone) with permission to download TOBI app from the Google Store or AppStore;
7. able to comply with outpatient clinic visits.

Exclusion Criteria:

* There are no exclusion criteria. All participants who meet inclusion criteria would be eligible to participate in the study.

Ages: 0 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 130 (Actual)
Dates: Start 2022-06-01 (Actual); Primary Completion 2024-03-08 (Actual); Study Completion 2024-03-08 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Medical University of South Carolina, Charleston, South Carolina, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Burn patients were recruited from burn clinic and the inpatient hospital setting to participate a study comparing face to face outpatient wound care to virtual wound care.
Pre-assignment Details: Parents/caregivers *and* children were considered enrolled in the study as a dyad, although most of the outcomes were reported by the parent instead of the child. Since demographic data was collected on both the caregiver and the child, the Total Started number is 130 (65 caregivers AND 65 children) as there were 65 dyads enrolled.
Groups:
- TOBI Arm: A novel smartphone application for burn wound care, called the Telemedicine Optimized Burn Intervention (TOBI), was developed to enable burn experts to direct burn wound care while the patient and caregiver are home through text messaging and video-conferencing. The app was designed to bring expert wound care directly to the patient's home to address barriers to healthcare, including high cost burden and time commitment (e.g., geographic limitations, transportation to burn centers, parking, lodging, meals, time away from school and work), particularly for patients/families in rural and medically underserved communities.
Period: Overall Study
Arm/Group | Face-to-face Arm | TOBI Arm
Started | 66 | 64
Caregivers | 33 | 32
Children | 33 | 32
Completed (For face-to-face 18 caregivers/18 children completed and for TOBI 21 caregivers/21 children completed the study.) | 36 | 42
Not Completed | 30 | 22

BASELINE CHARACTERISTICS:
Population: Parents/caregivers and patients were considered to be enrolled so baseline characteristics will be listed for both patients and their caregivers.
Groups:
- TOBI Arm: A novel smartphone application for burn wound care, called the Telemedicine Optimized Burn Intervention (TOBI), was recently developed to enable burn experts to direct burn wound care while the patient and caregiver are home through text messaging and video-conferencing. TOBI is synced with a portal used by providers, as an adjunct to standard therapy. This burn app provides education through frequently asked questions, instructional burn dressing change videos in addition to direct communication between patient and burn expert through store-and-forward pictures and videoconferencing.
  Telemedicine enhanced burn care: Participants assigned to TOBI will be given instructions how to download and use TOBI on a smartphone, including how to interface with burn clinicians using text-messaging, videoconferencing, and sending photos of the child's burn(s). The participants will have scheduled video visits with the care provider at least weekly until the burn has healed. The participants will be able to use other features of the app, such as text-messaging and sending photos of the burn(s), as needed. The participants will be able to use standard FTF burn care as well. They will be given instructions how to contact the burn team through the hospital paging operator if TOBI is unavailable or there is an emergency.
- Total: Total of all reporting groups
Arm/Group | Face-to-face Arm | TOBI Arm | Total
Number analyzed (Participants) | 66 | 64 | 130
Age, Categorical [Count of Participants; unit: Participants] — Population: Parents/caregivers and patients were considered to be enrolled so baseline characteristics will be listed for both patients and their caregivers.
  Participants
    Parents/Caregivers: number analyzed (Participants) | 33 | 32 | 65
    Parents/Caregivers: <=18 years | 0 | 0 | 0
    Parents/Caregivers: Between 18 and 65 years | 33 | 32 | 65
    Parents/Caregivers: >=65 years | 0 | 0 | 0
    Patients: number analyzed (Participants) | 33 | 32 | 65
    Patients: <=18 years | 33 | 32 | 65
    Patients: Between 18 and 65 years | 0 | 0 | 0
    Patients: >=65 years | 0 | 0 | 0
Age, Continuous [Median (Inter-Quartile Range); unit: years] — Population: Parents/caregivers and patients were considered to be enrolled so baseline characteristics will be listed for both patients and their caregivers.
  years
    Parents/Caregivers: number analyzed (Participants) | 33 | 32 | 65
    Parents/Caregivers | 34 [23.2 to 44.8] | 35 [25.2 to 44.8] | 34 [23 to 45]
    Patients: number analyzed (Participants) | 33 | 32 | 65
    Patients | 5 [1 to 8] | 8 [2.25 to 15] | 6 [1 to 10]
Sex: Female, Male [Count of Participants; unit: Participants] — Population: Parents/caregivers and patients were considered to be enrolled so baseline characteristics will be listed for both patients and their caregivers.
  Participants
    Parents/Caregivers: number analyzed (Participants) | 33 | 32 | 65
    Parents/Caregivers: Female | 28 | 32 | 60
    Parents/Caregivers: Male | 5 | 0 | 5
    Patients: number analyzed (Participants) | 33 | 32 | 65
    Patients: Female | 15 | 16 | 31
    Patients: Male | 18 | 16 | 34
Race (NIH/OMB) [Count of Participants; unit: Participants] — Population: Parents/caregivers and patients were considered to be enrolled so baseline characteristics will be listed for both patients and their caregivers.
  Participants
    Parents/Caregivers: number analyzed (Participants) | 33 | 32 | 65
    Parents/Caregivers: American Indian or Alaska Native | 0 | 0 | 0
    Parents/Caregivers: Asian | 0 | 0 | 0
    Parents/Caregivers: Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
    Parents/Caregivers: Black or African American | 13 | 13 | 26
    Parents/Caregivers: White | 15 | 18 | 33
    Parents/Caregivers: More than one race | 0 | 0 | 0
    Parents/Caregivers: Unknown or Not Reported | 5 | 1 | 6
    Patients: number analyzed (Participants) | 33 | 32 | 65
    Patients: American Indian or Alaska Native | 0 | 0 | 0
    Patients: Asian | 0 | 0 | 0
    Patients: Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
    Patients: Black or African American | 13 | 13 | 26
    Patients: White | 15 | 18 | 33
    Patients: More than one race | 0 | 0 | 0
    Patients: Unknown or Not Reported | 5 | 1 | 6
Region of Enrollment [Number; unit: participants]
  United States | 66 | 64 | 130

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Who Agree to Participate in the Study
Description: Looking at the number of participants (parents and children) who agree to enroll in the study at the time of burn injury versus the total number of participants who were approached to participate in the study.
Time Frame: At enrollment
Population: This includes caregivers and their children.
Measure: Number; unit: participants
Arm/Group | Face-to-face Arm | TOBI Arm
Number analyzed (Participants) | 84 | 72
participants | 66 | 64

2. Primary Outcome: Number of Participants Retained in the Study Over Time
Description: Looking at the number of participants retained in the study versus those lost to attrition
Time Frame: From enrollment to 30 days after burn wound has healed (up to 35 days after enrollment).
Population: Parents/caregivers and patients were considered to be enrolled together as a dyad, but are reported here as caregiver and patient.
Measure: Number; unit: participants
Groups:
- TOBI Arm: A novel smartphone application for burn wound care, called the Telemedicine Optimized Burn Intervention (TOBI), was recently developed to enable burn experts to direct burn wound care while the patient and caregiver are home through text messaging and video-conferencing. The app was designed to bring expert wound care directly to the patient's home to address barriers to healthcare, including high cost burden and time commitment (e.g., geographic limitations, transportation to burn centers, parking, lodging, meals, time away from school and work), particularly for patients/families in rural and medically underserved communities.
Arm/Group | Face-to-face Arm | TOBI Arm
Number analyzed (Participants) | 66 | 64
participants | 36 | 42

3. Primary Outcome: Wound Care Treatment Adherence
Description: Looking at the percentage of patient/caregiver dyads who adhered to prescribed burn wound care treatment protocol. A wound care fidelity checklist was used at each visit to determine the percentage of wound care adherence per visit. These percentages were then averaged for each weekly visit to give the value below.
Time Frame: Assessed weekly at clinic/telemedicine visit until burn wound was healed, up to 35 days after injury
Measure: Mean (Standard Deviation); unit: percentage of wound care adherence
Arm/Group | Face-to-face Arm | TOBI Arm
Number analyzed (Participants) | 66 | 64
percentage of wound care adherence | 76.8 (40.1) | 84.9 (29.1)

4. Primary Outcome: Number of Child Participants That Experienced Adverse Events, Serious Adverse Events, and Unexpected Problems
Description: Looking at the number of child participants in each condition that experienced adverse events, serious adverse events, and unexpected problems. Adverse events in this study included infection, delay in wound care or non-healing wound. Adult caregivers are not included in this as they did not have burn wounds that were assesssed.
Time Frame: Assessed weekly until burn wound was healed, up to 35 days
Measure: Count of Participants; unit: Participants
Arm/Group | Face-to-face Arm | TOBI Arm
Number analyzed (Participants) | 33 | 32
Participants | 0 | 0

5. Primary Outcome: Number of Times Problems With Technology Happened in the TOBI Condition
Description: Looking at the number of times providers or participants experienced and reported technological problems with TOBI
Time Frame: Assessed weekly until burn wound was healed, up to 35 days
Population: Only participants in the TOBI arm were evaluated for issues with technology as the face to face group did not interact with technology.
Measure: Number; unit: number of technological problems
Arm/Group | Face-to-face Arm | TOBI Arm
Number analyzed (Participants) | 0 | 64
number of technological problems |  | 1

6. Secondary Outcome: Number of Days Until Wound is Healed
Description: Looking at the number of days it takes for wound to heal following burn injury in both conditions
Time Frame: Measured during the treatment phase (2-4 weeks)
Measure: Mean (Standard Deviation); unit: days to wound healed
Arm/Group | Face-to-face Arm | TOBI Arm
Number analyzed (Participants) | 33 | 32
days to wound healed | 11.5 (4.3) | 11.4 (3.9)

7. Secondary Outcome: Number of Unscheduled ED or Clinic Visits
Description: Looking at the number of times participants had unscheduled visits (in the ED or the clinic)
Time Frame: Measured during the treatment phase (2-4 weeks)
Measure: Number; unit: number of unscheduled ED/clinic visits
Arm/Group | Face-to-face Arm | TOBI Arm
Number analyzed (Participants) | 33 | 32
number of unscheduled ED/clinic visits | 0 | 2

8. Secondary Outcome: Number of Wound Complications
Description: Looking at the number of wound complications (e.g., infection, conversion to deeper burn requiring surgery, conversion to deeper burn requiring a change in therapy).
Time Frame: Measured during the treatment phase (2-4 weeks)
Measure: Number; unit: number of wound complications
Arm/Group | Face-to-face Arm | TOBI Arm
Number analyzed (Participants) | 33 | 32
number of wound complications | 0 | 0

9. Secondary Outcome: Patient-reported Pain Scores
Description: Looking at average pain score at follow up visits between the two groups using the Wong-Baker Scale (0-10, with higher scores = more pain). Most patients only attended one follow up visit but if more than one, the average score is reported below.
Time Frame: Measured during the treatment phase (week 1 clinic visit)
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Face-to-face Arm | TOBI Arm
Number analyzed (Participants) | 33 | 32
units on a scale | 3.1 (3) | 1.8 (1.7)

10. Secondary Outcome: Caregiver's Perception of Child's Pain Scores
Description: Looking at average caregiver's perception of child's pain score at follow up visits between the two groups using the Wong-Baker Scale (0-10, with higher scores = more pain). Most dyads only attended one follow up visit but if more than one, the average score is reported below.
Time Frame: Measured during the treatment phase (week 1 clinic visit)
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Face-to-face Arm | TOBI Arm
Number analyzed (Participants) | 33 | 32
score on a scale | 3.1 (3.0) | 1.8 (1.7)

11. Secondary Outcome: Attitudes Towards Technology and Telemedicine Questionnaire
Description: Looking at the change in group average scores on the Attitudes Towards Technology and Telemedicine Questionnaire (caregiver-reported) from baseline to 1 month follow-up. Scores may range between 26-130, with higher scores = more positive attitudes towards technology and telemedicine.
Time Frame: Measured at baseline and 1-month follow-up
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Face-to-face Arm | TOBI Arm
Number analyzed (Participants) | 33 | 32
units on a scale | 79.5 (6.3) | 78.0 (8.4)

12. Secondary Outcome: Perception of Healthcare Access
Description: Looking at the change in group average scores on the Barriers to Care Questionnaire (BCQ), Pragmatics Subscale (caregiver-reported). Scores range from 0-100, with higher scores = fewer barriers and problems with access.
Time Frame: Measured at baseline and 1-month follow-up
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Face-to-face Arm | TOBI Arm
Number analyzed (Participants) | 31 | 32
units on a scale | 64.5 (25.5) | 72.6 (20.3)

13. Secondary Outcome: Positive And Negative Affect Schedule (PANAS) Scores
Description: Looking at the group average scores on the PANAS questionnaire measuring positive and negative affect (caregiver-reported). The means of the positive and negative scores for PANAS are reported below along with standard deviations. The scores range between 10-50, with higher scores = higher levels of affect (both positive and negative). For positive affect, a higher score is a better outcome and for negative affect, a lower score is a better outcome. Scores are reported for baseline and 1 month after burn wound healing.
Time Frame: Measured at baseline/enrollment and 1-month follow-up.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Face-to-face Arm | TOBI Arm
Number analyzed (Participants) | 31 | 32
units on a scale
  Baseline Positive Affect | 37 (7) | 32 (8)
  Baseline Negative Affect | 14 (4) | 13 (5)
  1 month follow up Positive Affect | 35 (8) | 33 (7)
  1 month follow up Negative Affect | 13 (4) | 11 (5)

14. Secondary Outcome: Patient-Reported Outcomes Measurement Information System - Depression (PROMIS-Depression) Scores
Description: Looking at the baseline and 1-month follow up scores on the Patient-Reported Outcomes Measurement Information System (PROMIS)-Depression questionnaire (caregiver-reported). Each item on the measure is rated on a 5-point scale (1=never; 2=rarely; 3=sometimes; 4=often; and 5=always) with a range in score from 8 to 40 with higher scores indicating greater severity of depression. The raw scores on the 8 items should be summed to obtain a total raw score. Next, the T-score table is used to identify the T-score associated with the individual's total raw score. The mean T-scores is 50 with a standard deviation of 10. T-scores range between 37.1-81.1. T scores are interpreted as follows: <55 (none to slight depression), 55-59.9 (mild depression), 60-69.9 (moderate depression), >70 (severe depression). T scores and standard error are reported below.
Time Frame: Measured at baseline and 1-month follow-up
Measure: Mean (Standard Error); unit: T-score
Arm/Group | Face-to-face Arm | TOBI Arm
Number analyzed (Participants) | 31 | 32
T-score
  Baseline | 47.5 (7.6) | 47.5 (6.2)
  1 month follow up | 47.5 (8.0) | 44.9 (6.1)

15. Secondary Outcome: Patient-Reported Outcomes Measurement Information System - Anxiety (PROMIS-Anxiety) Scores
Description: Looking at the baseline and 1-month follow up scores on the Patient-Reported Outcomes Measurement Information System (PROMIS)-Anxiety questionnaire (caregiver-reported). Each item on the measure is rated on a 5-point scale (1=never; 2=rarely; 3=sometimes; 4=often; and 5=always) range in score from 7 to 35 with higher scores indicating greater severity of anxiety. The raw scores on the 7 items should be summed to obtain a total raw score. Next, the T-score table is used to identify the T-score associated with the individual's total raw score. The mean T-scores is 50 with a standard deviation of 10. T-scores range between 36.3-82.7. T scores are interpreted as follows: <55 (none to slight anxiety), 55-59.9 (mild anxiety), 60-69.9 (moderate anxiety), >70 (severe anxiety). T scores and standard error are reported below.
Time Frame: Measured at baseline and 1-month follow-up
Measure: Mean (Standard Error); unit: T-score
Arm/Group | Face-to-face Arm | TOBI Arm
Number analyzed (Participants) | 31 | 32
T-score
  Baseline | 50.7 (9.1) | 47.8 (7.8)
  1 month follow up | 50.4 (6.8) | 46.8 (7.6)

16. Secondary Outcome: Patient-Reported Outcomes Measurement Information System - General Self-Efficacy (PROMIS-General-Self-Efficacy) Scores
Description: Looking at the baseline and 1-month follow up scores on the Patient-Reported Outcomes Measurement Information System (PROMIS)-General Self Efficacy questionnaire (caregiver-reported). Each item on the measure is rated on a 5-point scale (1=never; 2=rarely; 3=sometimes; 4=often; and 5=always) range in score from 8 to 40 with higher scores indicating greater self efficacy. The raw scores on the 7 items should be summed to obtain a total raw score. Next, the T-score table is used to identify the T-score associated with the individual's total raw score. The mean T-scores is 50 with a standard deviation of 10. T-scores range between 22.72-64.98. A T-score value of 55 indicated that the respondent has greater self-efficacy for managing emotions. Higher scores indicating more self efficacy and lower scores with less self efficacy. T scores and standard error are reported below.
Time Frame: Measured at baseline only
Measure: Mean (Standard Error); unit: T-score
Arm/Group | Face-to-face Arm | TOBI Arm
Number analyzed (Participants) | 31 | 32
T-score | 53.5 (10.1) | 53.2 (8.8)

17. Secondary Outcome: Patient-Reported Outcomes Measurement Information System - Self-Efficacy to Manage Emotions (PROMIS-Self-Efficacy-Manage-Emotions) Scores
Description: Looking at the baseline and 1-month follow up scores on the Patient-Reported Outcomes Measurement Information System (PROMIS)-Self-Efficacy Managing emotions questionnaire (caregiver-reported). Each item on the measure is rated on a 5-point scale (1=never; 2=rarely; 3=sometimes; 4=often; and 5=always) range in score from 4-20 with higher scores indicating greater severity of anxiety. The raw scores on the 4 items should be summed to obtain a total raw score. Next, the T-score table is used to identify the T-score associated with the individual's total raw score. The mean T-scores is 50 with a standard deviation of 10. T-scores range between 36.3-82.7. A T-score of 55 and greater indicates that the respondent has greater self efficacy and ability to manage their emotions regarding disease. A higher score than 55 indicates even more self efficacy and lower score, less. T scores and standard error are reported below.
Time Frame: Measured at baseline only
Measure: Mean (Standard Error); unit: T-score
Arm/Group | Face-to-face Arm | TOBI Arm
Number analyzed (Participants) | 31 | 32
T-score | 50.2 (9.1) | 50.7 (6.6)

18. Secondary Outcome: Peritraumatic Distress Inventory (PDI) Sores
Description: Looking at average scores on the Peritraumatic Distress Inventory (caregiver-reported). Scores range between 0-52, with higher scores = greater peritraumatic distress. An optimal cutoff score of 23 (sensitivity = 71%; specificity = 73%) is good for predicting clinically elevated PTSD 30-days post-injury.
Time Frame: Measured at baseline only
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Face-to-face Arm | TOBI Arm
Number analyzed (Participants) | 31 | 32
units on a scale | 11.9 (8.1) | 13.8 (8.3)

19. Secondary Outcome: Perceived Stress Scale (PSS) Scores
Description: Looking at average scores on the Perceived Stress Scale (caregiver-reported) between two conditions. Scores on the PSS can range from 0 to 40 with higher scores = higher perceived stress. Scores ranging from 0-13 would be considered low stress. Scores ranging from 14-26 would be considered moderate stress. Scores ranging from 27-40 would be considered high perceived stress.
Time Frame: Measured at 1-month follow-up only
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Face-to-face Arm | TOBI Arm
Number analyzed (Participants) | 31 | 32
units on a scale | 18.6 (2.7) | 19.4 (3.0)

20. Secondary Outcome: Posttraumatic Growth Inventory (PTGI) Scores
Description: Average scores on the Posttraumatic Growth Inventory (caregiver-reported). Scores range from 0-105, with higher scores = greater posttraumatic growth.
Time Frame: Measured at 1-month follow-up only
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Face-to-face Arm | TOBI Arm
Number analyzed (Participants) | 31 | 32
units on a scale | 54.7 (31.9) | 39.5 (35.6)

21. Secondary Outcome: Client Satisfaction Questionnaire-8 (CSQ-8) Scores
Description: Looking at average scores on the Client Satisfaction Questionnaire-8 scores (caregiver-reported). Scores range between 8-32, with higher scores = greater satisfaction.
Time Frame: Measured at 1-month follow-up only
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Face-to-face Arm | TOBI Arm
Number analyzed (Participants) | 31 | 32
units on a scale | 30.8 (3) | 30.5 (3)

22. Secondary Outcome: mHealth App Usability Questionnaire (MAUQ) Scores
Description: Looking at average scores on the MAUQ questionnaire measuring app usability (caregiver-reported in TOBI condition only). Raw scores range between 21-147 and average scores range between 1-7, with higher overall score equivalent to higher usability of the app. The average scores and standard deviation are reported below for the TOBI group.
Time Frame: Measured at 1-month follow-up only
Population: The face-to-face arm did not use the TOBI app at all, therefore they did not take the MAUQ to rate the app.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Face-to-face Arm | TOBI Arm
Number analyzed (Participants) | 0 | 32
units on a scale |  | 6.3 (0.8)

23. Secondary Outcome: Total Number of Face-to-face Visits
Description: Looking at the total number of face-to-face visits
Time Frame: Treatment phase (weeks 2-4)
Measure: Mean (Standard Deviation); unit: number of visits
Arm/Group | Face-to-face Arm | TOBI Arm
Number analyzed (Participants) | 66 | 64
number of visits | 2.1 (0.8) | 1.1 (0.3)

24. Secondary Outcome: Total Number of TOBI Visits
Description: Looking at the total number of TOBI visits
Time Frame: Treatment phase (weeks 2-4)
Population: This outcome only pertains to the TOBI arm as the face-to-face arm did not have any TOBI visits.
Measure: Mean (Standard Deviation); unit: number of visits
Arm/Group | Face-to-face Arm | TOBI Arm
Number analyzed (Participants) | 0 | 64
number of visits |  | 1.1 (0.6)

25. Secondary Outcome: Total Travel Time
Description: Looking at the total travel time in each condition as reported by the caregiver.
Time Frame: From enrollment through treatment phase (weeks 1-4)
Measure: Mean (Standard Deviation); unit: hours
Arm/Group | Face-to-face Arm | TOBI Arm
Number analyzed (Participants) | 33 | 32
hours | 4.0 (3.1) | 2.3 (2.5)

26. Secondary Outcome: Direct Cost to Patient/Caregiver
Description: Looking at the direct cost to patient/caregiver as reported by caregiver
Time Frame: From enrollment through treatment phase (weeks 1-4)
Measure: Mean (Standard Deviation); unit: dollars
Arm/Group | Face-to-face Arm | TOBI Arm
Number analyzed (Participants) | 33 | 32
dollars | 339.10 (568.14) | 258.81 (390.38)

27. Secondary Outcome: Time to Return to Work
Description: Looking at the average time it took patient/caregiver to return to work after burn wound injury.
Time Frame: From enrollment through the treatment phase (weeks 1-4). This included any time that the parent had was out of work because of the injury at time of occurrence or due to clinic follow up.
Measure: Mean (Standard Deviation); unit: days
Arm/Group | Face-to-face Arm | TOBI Arm
Number analyzed (Participants) | 33 | 32
days | 2.0 (2.2) | 1.3 (1.5)

ADVERSE EVENTS:
Time Frame: For each child participant dyad, adverse event data was only collected on the child participant up to 46 days after burn wound injury.
Description: Adult participants of the dyad were not monitored for adverse events as they did not have burn injuries and are not reported here.
Arm/Group | Face-to-face Arm | TOBI Arm
All-Cause Mortality (participants affected / at risk) | 0/33 | 0/32
Serious Adverse Events (participants affected / at risk) | 0/33 | 0/32
Other Adverse Events (participants affected / at risk) | 0/33 | 2/32
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Face-to-face Arm (N=33) | TOBI Arm (N=32)
Unscheduled visit to the ED or Clinic (Skin and subcutaneous tissue disorders) | 0 (0) | 2 (2) — In either arm, we tracked the number of unscheduled or unplanned patient visits to the ED or clinic.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2023-07-01): https://cdn.clinicaltrials.gov/large-docs/44/NCT05019144/Prot_SAP_001.pdf
  • Informed Consent Form (2022-07-26): https://cdn.clinicaltrials.gov/large-docs/44/NCT05019144/ICF_000.pdf